CLINICAL TRIAL: NCT02875431
Title: Registry for the Detection of C5 Palsy After ACDF
Brief Title: Multicentric Registry for the Detection of C5 Palsy After Anterior Cervical Discectomy and Fusion
Acronym: C5registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Collaborators: Medical University Innsbruck (Other); Charite University, Berlin, Germany (Other); University Hospital, Geneva (Other); Klinik für Neurochirurgie, Köln-Mehrheim (Unknown); Wirbelsäulenzentrum, St. Josephs-Hospital, Wiesbaden (Unknown); Vivantes Clinic Neukölln (Other); Klinik für Neurochirurgie, Helios-Klinikum Krefeld (Unknown); Universitätsklinikum Hamburg-Eppendorf (Other); Klinikum Karlsbad-Langensteinbach (Other); Ludwig-Maximilians - University of Munich (Other); Zentrum für Wirbelsäulenchirurgie Kempen (Unknown)
Responsible Party: Sponsor
Other Study IDs: C5 registry
Record Dates: First submitted 2016-08-12; First posted 2016-08-23 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Degenerative Cervical Spinal Stenosis; Cervical Disc Herniation; Suspected Cervical Spine Instability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ACDF or cervical vertebral body replacement
  Interventions: Procedure: Patients undergo ACDF or cervical vertebral body replacement

INTERVENTIONS:
Procedure: Patients undergo ACDF or cervical vertebral body replacement

SUMMARY:
Detect the reason for the frequently occurring C5 palsy after anterior cervical discectomy and fusion

DETAILED DESCRIPTION:
A registry which includes all known and individually analyzed but even new factors are evaluated in order to perform a multivariate analysis for the detection of risk factors of C5 palsy after anterior cervical discectomy and fusion which is a very disabling and still cryptic complication.

ELIGIBILITY:
Inclusion Criteria:

* ACDF or cervical vertebral body replacement due to herniated disc, spinal stenosis or trauma

Exclusion Criteria:

* infectious disease or neurodegenerative disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ACDF or cervical vertebral body replacement due to herniated disc, spinal stenosis or trauma
Sampling Method: Non-Probability Sample
Enrollment: 1087 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
C5 palsy | 3 months
  defined as deterioration on BMRC scale of C5 innervated muscles

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Meyer, MD, Study Chair — TU München
Locations (1):
- Department of Neurosurgery, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No